CLINICAL TRIAL: NCT05876195
Title: Varying Keyhole Limpet Haemocyanin-adjuvant Dose Combinations to Explore the Immune Response: a Human Challenge Study
Brief Title: KLH Challenge to Explore the Human Immune Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16114
Record Dates: First submitted 2023-03-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-03

CONDITIONS: Immune Response
Keywords: Keyhole Limpet Hemocyanin; Keyhole Limpet Haemocyanin; KLH; Human immune challenge; Proof of mechanism; Experimental Medicine; Adjuvant; Montanide; Alhydrogel
MeSH Terms: interventions — keyhole-limpet hemocyanin; Sodium Chloride; Saline Solution; montanide ISA 51; Aluminum Hydroxide

STUDY DESIGN:
Intervention Model Description: Parallel group randomised experimental medicine study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1: Saline 0.9% (placebo) primary dose (Placebo Comparator): IM saline 0.9% (placebo) day 0, followed by multi-dose ID subunit KLH (0 mcg (saline), 1 mcg, 3 mcg, 10mcg, 30mcg, 100mcg) day 28
  Interventions: Drug: Saline
- Group 2: subunit KLH 1000mcg primary dose (Active Comparator): IM dose subunit KLH 1000 mcg day 0, followed by multi-dose ID subunit KLH (0 mcg (saline), 1 mcg, 3 mcg, 10mcg, 30mcg, 100mcg) day 28
  Interventions: Biological: Keyhole-Limpet Hemocyanin
- Group 3: subunit KLH 1000mcg plus aluminium hydroxide adjuvant 900mcg primary dose (Active Comparator): IM dose subunit KLH 1000 mcg plus aluminium hydroxide 900mcg day 0, followed by multi-dose ID subunit KLH (0 mcg (saline), 1 mcg, 3 mcg, 10mcg, 30mcg, 100mcg) day 28
  Interventions: Biological: Keyhole-Limpet Hemocyanin; Drug: Alhydrogel
- Group 4: subunit KLH 1000mcg plus Montanide ISA-51 primary dose (Active Comparator): IM dose subunit KLH 1000 mcg plus Montanide ISA-51 day 0, followed by multi-dose ID subunit KLH (0 mcg (saline), 1 mcg, 3 mcg, 10mcg, 30mcg, 100mcg) day 28
  Interventions: Biological: Keyhole-Limpet Hemocyanin; Drug: Montanide ISA 51 VG
- Group 5: subunit KLH 10mcg primary dose (Active Comparator): IM dose subunit KLH 10 mcg day 0, followed by multi-dose ID subunit KLH (0 mcg (saline), 1 mcg, 3 mcg, 10mcg, 30mcg, 100mcg) day 28
  Interventions: Biological: Keyhole-Limpet Hemocyanin
- Group 6: subunit KLH 10mcg plus aluminium hydroxide adjuvant 900mcg primary dose (Active Comparator): IM dose subunit KLH 10 mcg plus aluminium hydroxide 900mcg day 0, followed by multi-dose ID subunit KLH (0 mcg (saline), 1 mcg, 3 mcg, 10mcg, 30mcg, 100mcg) day 28
  Interventions: Biological: Keyhole-Limpet Hemocyanin; Drug: Alhydrogel
- Group 7: subunit KLH 10mcg plus Montanide ISA-51 primary dose (Active Comparator): IM dose subunit KLH 10 mcg plus Montanide ISA-51 day 0, followed by multi-dose ID subunit KLH (0 mcg (saline), 1 mcg, 3 mcg, 10mcg, 30mcg, 100mcg) day 28
  Interventions: Biological: Keyhole-Limpet Hemocyanin; Drug: Montanide ISA 51 VG
- Group 8: Blood-sample only group (non-randomised) (No Intervention): No challenge agent, blood sampling only.

INTERVENTIONS:
Biological: Keyhole-Limpet Hemocyanin — Sub-unit Keyhole Limpet Haemocyanin (KLH, Immucothel, Biosyn, Fellbach, Germany)
  Other Names: KLH; Immucothel
  Arms: Group 2: subunit KLH 1000mcg primary dose; Group 3: subunit KLH 1000mcg plus aluminium hydroxide adjuvant 900mcg primary dose; Group 4: subunit KLH 1000mcg plus Montanide ISA-51 primary dose; Group 5: subunit KLH 10mcg primary dose; Group 6: subunit KLH 10mcg plus aluminium hydroxide adjuvant 900mcg primary dose; Group 7: subunit KLH 10mcg plus Montanide ISA-51 primary dose
Drug: Saline — Placebo intervention.
  Other Names: Normal saline; 0.9% Saline
  Arms: Group 1: Saline 0.9% (placebo) primary dose
Drug: Montanide ISA 51 VG — Montanide ISA-51 (Seppic, France) is a water-in-oil vaccine adjuvant
  Other Names: Montanide ISA 51
  Arms: Group 4: subunit KLH 1000mcg plus Montanide ISA-51 primary dose; Group 7: subunit KLH 10mcg plus Montanide ISA-51 primary dose
Drug: Alhydrogel — Alhydrogel is a vaccine adjuvant
  Other Names: Aluminum hydroxide adjuvant 2%
  Arms: Group 3: subunit KLH 1000mcg plus aluminium hydroxide adjuvant 900mcg primary dose; Group 6: subunit KLH 10mcg plus aluminium hydroxide adjuvant 900mcg primary dose

SUMMARY:
One approach to improve the efficiency of the drug development process is the use of human 'immune challenge' studies. In these studies, healthy volunteers are given small amounts of substances which are foreign to their immune system to provoke a temporary response: the 'challenge'. Depending on the nature and dose of the challenge, the body's immune system will react in a different but predictable way, elements of which mimic those seen in disease, thereby 'modelling' them. These models can help safely bridge the gap between animal experiments and patient groups and, if sufficiently understood, test the effect of new drugs without exposing patients to risk. Sadly, whilst immune challenge models have been used in drug development for many years, this has been done in a largely non-standardised, ad hoc manner, which greatly limits the usefulness of the approach.

The purpose of this research is to better understand, improve, and standardise a common method of immune challenge which uses a protein called 'Keyhole Limpet Haemocyanin' (KLH). KLH is available as a highly-purified formulation, and because it is not usually encountered by the human immune system (it is derived from an inedible shellfish), it allows us to study the development of immune responses right from the time it is administered. We plan to give different groups of healthy volunteers different doses of KLH with or without an 'immune-boosting' agent (Alhydrogel™ or Montanide ISA™51, commonly referred to as adjuvants), before measuring and comparing their response. We will then re-challenge all the volunteers a month later by injecting different doses of KLH into the skin on their forearms, similar to an allergy test, taking images, blood samples and skin biopsies to understand the nature, time course, and variability of the immune response in each individual. No previous studies have directly explored the effects of KLH dose or adjuvants in a rigorous manner. The results will help us to determine both whether administering KLH with different adjuvants elicits qualitatively different immune response profiles (thus modelling different diseases) and the optimal doses of KLH to evaluate new drugs with. In turn, we hope this will help improve the percentage of drugs progressing from concept to clinical therapy, addressing unmet health needs.

DETAILED DESCRIPTION:
This is a single blind, parallel group, two-phase challenge study to determine the relative immunogenicity of subunit KLH, with and without aluminium hydroxide adjuvant, in healthy UK volunteers aged 18-45. The prime dose of subunit KLH (+/- aluminium hydroxide or Montanide ISA-51) will be administered IM, and the re-challenge dose of subunit KLH for assessment of DTH will be administered ID.

This trial will be conducted at a Clinical Research Facility based at the University of Oxford supporting researchers from Oxford University Joint Research Office (JRO) approved research.

There will be 7 randomised study groups (plus one non-randomised 'blood sample only' group, group 8 - see section 8.6) and it is anticipated that a maximum of 39 volunteers will be enrolled (excluding dropouts). Eligible participants will be randomised into any of 7 study groups (section 7.1) according to study phase. Randomisation and enrolment will occur in two phases. Phase 1 will consist of group 1 (placebo prime dose) and the standard (1000mcg) KLH dose +/- adjuvant groups (2, 3, and 4). Following interim analysis of data from these 21 participants, recruitment into Phase 2 (the lower [10mcg] KLH dose groups: groups 5,6,7) will occur provided there is sufficient evidence of immunogenicity in the standard dose group.

Should participants withdraw or dropout of the study, replacement volunteers will be enrolled to ensure the target number of participants per group is achieved with all participants competing the full follow-up period. A maximum of 6 additional volunteers may be sought for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study and is able to comply with the study protocol.
* Male or female between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a physician, based on a detailed medical history and a complete physical examination including vital signs and laboratory measurements.
* Body weight >= 50 kg and body mass index (BMI) within the range 18 to 30 kilogram/meter squared (inclusive).
* Female participants of child bearing potential: Females of child bearing potential are eligible to enter if they are not pregnant (negative pregnancy test on the day of both screening and vaccination) and willing to use effective methods of contraception to prevent pregnancy from the time of first dose to 60 days afterwards.
* Male participants with female partners of child-bearing potential: must agree to use effective methods of contraception from the time of the first dose of challenge agent to 60 days afterwards.
* At least 2 previous doses of a registered SARS-CoV2 vaccination, at least 60 days previously
* Sufficient English language ability to enable appropriate informed consent procedures to be conducted in English

Exclusion Criteria:

* Antibiotics or antiviral therapy after a serious illness within 30 days of study entry.
* SARS CoV2 (COVID-19) infection within the previous 30 days, diagnosed using PCR test or lateral flow device
* Any use of immunosuppressant or immunomodulatory agents (systemic or topical) in 3 months prior to study entry.
* Chronic medical conditions with potential effect on immune responses including diabetes, significant history of atopy, or any condition that, in the opinion of the investigator, would interfere with the study
* Presence of tattoos, naevi or other skin abnormalities such as keloids (or history of keloids) that may, in the opinion of the investigator, interfere with study assessments.
* Fitzpatrick skin type V and VI (due to potential interference with assessment of DTH response)
* Pregnancy or breastfeeding
* Allergy to KLH, aluminium hydroxide, Montanide ISA-51, related vaccine adjuvants, or components of the study challenge agents
* Allergy to shellfish
* Residency in or significant previous travel to areas endemic for schistosomiasis (due to potential cross-reactive immune responses to KLH)
* Previous exposure to Keyhole Limpet Haemocyanin, e.g. in the context of a previous study
* Participants participating, within 7 days of screening, in recreational sun-bathing, or use of sun-bed, on the area of the skin from wrist to shoulder inclusive.
* Phobia of needles or minor surgical procedures.
* Current smoker or using nicotine replacement therapy
* Participants receiving any vaccinations within 2 months prior to screening visit, or will require vaccination prior to the end of study follow-up.
* Any other significant disease, disorder, or finding, which, in the opinion of the investigator, may either put the participant at risk, affect their ability to participate in the study or impair interpretation of the study data

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
To establish the immunogenicity of subunit KLH at different doses, with and without aluminium hydroxide or Montanide ISA-51 adjuvants | Day 28
  Proportion of participants with >2-fold increase over baseline (D0) in anti-KLH IgG antibody titre by ELISA in each group

SECONDARY OUTCOMES:
Determine whether different doses of subunit KLH, with and without aluminium hydroxide or Montanide ISA-51 adjuvants, elicit predominantly TH1, TH2 or balanced responses | Day 28
  Ratio of TH1:TH2 antigen responsive cells based on number of IFN- γ (TH1) and IL-4 (TH2) producing PBMCs (cells per 10^6 PBMC) in response to KLH stimulation by ELISpot in each group.
Within-participant dose-response to intradermal KLH on day Day 28: skin induration response (EC50) | Day 30 (48 hours after Day 28 KLH re-challenge)
  Intradermal KLH dose required for 50 percent of maximal induration response (EC50, measured in mm)
Within-participant dose-response to intradermal KLH on day Day 28: skin induration response (Emax) | Day 30 (48 hours after Day 28 KLH re-challenge)
  Maximal induration response to intradermal KLH dose (Emax, measured in mm)
Within-participant dose-response to intradermal KLH on day Day 28: skin erythema response (EC50) | Day 30 (48 hours after Day 28 KLH re-challenge)
  Intradermal KLH dose required for 50 percent of maximal erythema response (EC50, measured in mm)
Within-participant dose-response to intradermal KLH on day Day 28: skin erythema response (Emax) | Day 30 (48 hours after Day 28 KLH re-challenge)
  Maximal erythema response to intradermal KLH dose (Emax, measured in mm)

CONTACTS AND LOCATIONS:
Overall Officials: James Fullerton, MBBS, Principal Investigator — NDORMS, University of Oxford
Locations (1):
- NIHR Oxford Experimental Medicine Clinical Research Facility, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only non-identifiable data anonymised to the ICO Anonymisation: managing data protection risk code of practice generated in this study will be suitable for sharing. We will adhere to the MRC's policy on data sharing.
  ORA-data offers a means for Oxford's researchers to openly share non-confidential research data, without the need for external data users to undergo authentication. Each deposit is accompanied by appropriate metadata and is assigned a unique Digital Object Identifier (DOI) via the DataCite scheme, allowing it to be cited in publications. Directions to key datasets will also be made available via the group's web page on the Institute's web site. Appropriate metadata will be published with research data to enable other researchers to identify whether the data could be suitable for their own research.
Time Frame: The study team will have exclusive use of the data for a reasonable period of time following the completion of the study in order to complete analysis and secure publication of results.
Access Criteria: As per MRC Policy and Guidance on Sharing of Research Data from Population and Patient Studies and the Oxford University Data Sharing Policy, any external users will be required to agree to terms set out in an Oxford University Data Sharing Agreement. The agreement will outline their responsibilities and will prohibit any attempt to identify study participants, breach confidentiality or make unapproved contact with study participants.
URL: http://www.bodleian.ox.ac.uk/bdlss/digital-services/data-archiving